CLINICAL TRIAL: NCT01119118
Title: Pharmacodynamic Response Assessment With PET/MRI Imaging in Patients With Metastatic Prostate CAncer to Bone Treated With ZD4054
Brief Title: ZD4054 With Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI) for Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO09805; NCI-2011-00736 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison); H-2009-0160 (Other: Institutional Review Board)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2013-04-29 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: Metastatic; castrate-resistant prostate cancer; bone metastasis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): ZD4054 + multimodal PET/MRI imaging
  Interventions: Drug: ZD4054

INTERVENTIONS:
Drug: ZD4054 — All patients will be treated with ZD4054 at 10 mg PO daily, repeated in four week cycles (1 cycle = 28 days). All patients will initially undergo NaF and FDG PET/CT and MRI imaging at baseline (scan#1), and then again after 4 weeks (scan#2) of ZD4054 exposure. Subsequently, ZD4054 will be held for 2 weeks followed by the final NaF and FDG-PET/CT and MRI acquisition (scan#3). After the final PET/MRI is obtained, patients will resume ZD4054 and be assessed for safety prior to each new cycle of therapy. Standard disease evaluation assessments will be conducted after cycle#3, and repeated after every third cycle (sooner if clinically indicated). Therapy will continue until radiographical/clinical disease progression or unacceptable toxicity

SUMMARY:
The purpose of this research study is to assess the effects of ZD4054 on prostate cancer that has spread to the bones by using new imaging techniques. In particular, this study will use fluorodeoxyglucose (FDG) and 18F-Sodium Fluoride (NaF) PET/computed tomography (CT) and MRI scans to look for changes in bone metastasis after ZD4054 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Men > 18 years of age.
2. Histologically proven adenocarcinoma of the prostate.
3. Presence of radiographic bone metastasis with at least one which is amenable to serial imaging using MRI/PET imaging.
4. Patients must have evidence of progressive disease by either radiographic progression or a rising PSA within 4 weeks prior to registration.
5. Patients must have had prior treatment with bilateral orchiectomy or other primary androgen-deprivation therapy.
6. For patients previously treated with flutamide (Eulexin), Nilutamide (Nilandron), or bicalutamide (Casodex): Patients must have discontinued flutamide > 4 weeks prior to registration with continued evidence of progressive disease. For bicalutamide or nilutamide, patients must have discontinued the drug > 6 weeks prior to registration with evidence of progressive disease.
7. Prior therapy is permitted as long as it was given > 4 weeks prior to registration, and evidence for disease progression is met.
8. Patients must not have had prior radiotherapy < 4 weeks prior to registration.
9. Prior use of bisphosphonates allowed only if started at least 12 or more weeks prior to registration (can continue current dose/schedule while on study).
10. Patient cannot have had prior Strontium 89, Samarium 153, or other radioisotope.
11. No concurrent use of estrogen, or estrogen-like agents
12. Patients must have adequate organ function
13. ECOG performance status 0-2.

Exclusion Criteria:

1. Use of potent CYP450 inducers (such as phenytoin, rifampicin, carbamazepine and phenobarbitone, St. John's Wort) within 2 weeks prior to start of study treatment.
2. Prior therapy with endothelin receptor antagonists or family history of hypersensitivity to endothelin antagonists.
3. History of past or current epilepsy, epilepsy syndrome, or other seizure disorder.
4. Stage II, III or IV cardiac failure (classified according to New York Heart Association (NYHA) classification), myocardial infarction within 6 months prior to study entry, or have left ventricular function (LVEF) below the institutional normal limit.
5. QT interval corrected for heart rate (by Bazett's correction) (QTcB) >470 msec.
6. Previous history or presence of another cancer, other than prostate cancer or treated squamous/basal cell carcinoma of the skin, within the last 5 years.
7. Major surgery within 6 weeks of registration.
8. Hemoglobin (Hb) <9 g/dL. Concomitant use of erythropoietin or blood transfusions is allowed.
9. Inability to take or absorb oral medications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Simoncic U, Perlman S, Liu G, Staab MJ, Straus JE, Jeraj R. Comparison of NaF and FDG PET/CT for assessment of treatment response in castration-resistant prostate cancers with osseous metastases. Clin Genitourin Cancer. 2015 Feb;13(1):e7-e17. doi: 10.1016/j.clgc.2014.07.001. Epub 2014 Jul 15. PMID 25128349
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at the University of Wisconsin Carbone Cancer Center from April 2010 until July 2011.
Groups:
- ZD4054: ZD4054 therapy at the starting dose of 10 mg PO with multimodal PET/MRI imaging
Period: Overall Study
Arm/Group | ZD4054
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- ZD4054: ZD4054 + multimodal PET/MRI imaging
Arm/Group | ZD4054
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6
Prior Therapy [Number; unit: Participants]
  Prior Antiandrogen and Cytotoxic Chemotherapy | 5
  Prior Antiandrogen Therapy (no prior chemo) | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Whose Tumor Lesion Size Changed After 6 Weeks of Treatment With ZD4054 Using PET and MRI Scans.
Description: Multimodal Positron Emission Tomography (PET) and Magnetic Resonant Imaging (MRI) imaging were used to evaluate changes in the tumor lesion size following 6 weeks of treatment with ZD4054.
Time Frame: Week 6
Measure: Number; unit: participants
Arm/Group | ZD4054
Number analyzed (Participants) | 6
participants | 0

2. Secondary Outcome: The Number of Subjects Whose Tumor Lesion Size Changed Using Positron Emission Tomography (PET) Imaging Alone.
Time Frame: Week 6
Measure: Number; unit: participants
Arm/Group | ZD4054
Number analyzed (Participants) | 6
participants | 0

3. Secondary Outcome: The Number of Subjects Whose Tumor Lesion Size Changed Using Diffusion-weighted Imaging (DWI)-Magnetic Resonant Imaging (MRI) Alone
Time Frame: Week 6
Measure: Number; unit: participants
Arm/Group | ZD4054
Number analyzed (Participants) | 6
participants | 0

4. Secondary Outcome: Number of Subjects Whose Tumor Lesion Size Changed Using Iterative Decomposition of Water and Fat With Echo Asymmetry and Least-squares Estimation (IDEAL)-MRI Imaging Alone
Time Frame: Week 6
Measure: Number; unit: participants
Arm/Group | ZD4054
Number analyzed (Participants) | 6
participants | 0

5. Secondary Outcome: Number of Subjects With PSA Response
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | ZD4054
Number analyzed (Participants) | 6
participants | 0

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | ZD4054
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZD4054 (N=6)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZD4054 (N=6)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Fever (General disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1 (1)
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bronchus (Infections and infestations) | 1 (1)
Edema: limb (General disorders) | 1 (1)
AST increased (Investigations) | 1 (1)
Albumin, serum-low (Investigations) | 1 (1)
Calcium, serum-low (hypocalcemia) (Investigations) | 1 (1)
Sodium, serum-low (hyponatremia) (Investigations) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Mood alteration - Depression (Psychiatric disorders) | 1 (1)
Neurology - Other (Psychiatric disorders) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Head/headache (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes